CLINICAL TRIAL: NCT00236210
Title: The Vascular Intervention Project (VIP): a Randomized Controlled Trial of a Novel Community-based Primary and Secondary Cardiovascular Prevention Program in the Algoma District of Northern Ontario
Brief Title: A Randomized Controlled Trial of a Novel Community-based Primary and Secondary Cardiovascular Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Group Health Centre (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); McMaster University (Other); Coalition for the Acquisition of Sound Habits (Other); Ministry of Northern Development and Mines Youth Internship Program (Unknown); Pfizer (Industry)
Responsible Party: Dr. David Crookston, Group Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Go3-03031
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-07

CONDITIONS: Vascular Disease; Diabetes; Hypertension; Hyperlipidemia; Obesity
Keywords: Vascular Intervention Program; Vascular Disease; Coronary Artery Disease; Diabetes; Lifestyle Modification; Modifiable Risk Factors
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Hypertension; Hyperlipidemias; Obesity; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIP program (Active Comparator): Risk assessment, lifestyle counselling, exercise program
  Interventions: Behavioral: Action Score; Behavioral: VIP program
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Action Score — Improvement in a novel 100-point score summarizing cardiovascular risk.
  Arms: VIP program
Behavioral: VIP program — Risk assessment, lifestyle counselling, exercise program
  Arms: VIP program

SUMMARY:
VIP is a demonstration project with a goal to decrease modifiable risk factors for those with a higher risk of having a vascular event such as a heart attack or stroke or of developing vascular disease. Introduced as a study, VIP compares whether there is a significant reduction of modifiable vascular risk factors among patients who are involved in a personalized directed program versus those being provided standard care by their physician. Health care providers work collaboratively with the 'VIP Team' to improve the participants' vascular health.

DETAILED DESCRIPTION:
This Northern Ontario, community-based demonstration project is a multi-disciplinary, primary care provider-based collaboration. The goals of the project are to:

1. Decrease the modifiable risk factors for primary care patients at risk for vascular disease in the Algoma District;
2. Increase collaboration between health care providers such as family physicians, pharmacists, physiotherapists, dietitians and nurses in the community;
3. Increase the participation of the patient and family in decision-making, self-care, and adherence to agreed-upon management plans;
4. Improve patient access to care, clinical outcomes and satisfaction;
5. Provide a business case for a practical, sustainable and generalizable model for the primary care of vascular disease in the community.

The Group Health Centre, a multi-disciplinary, not-for-profit community-based health organization with 56,000 rostered patients, leads the project. However, all Sault Ste Marie community patients are eligible to join the Vascular Intervention Program (VIP). This program has three key components: a registry of VIP patients with audit, recall and feedback; use of the novel ACTION score template, and the optional use of VIPNet, a personalized patient record tool that provides secure web access to optimize quality and continuity of care. The VIP project aims to empower patients and increase collaboration among the primary health care team. Patients with any vascular risk factors will be eligible for VIP.

The VIP project is a demonstration project that does not duplicate existing GHC chronic disease management programs because (1) the VIP is offered to all eligible community patients, not only GHC enrollees; (2) VIP integrates any patients with vascular risk, not just those with pre-defined conditions; (3) novel collaborative tools such as the ACTION template and VIPNet website are being piloted; and (4) explicit patient-centred decision making drives the process. The development and evaluation of the VIP demonstration project is a unique step in the evolution of primary care chronic disease management in Sault Ste Marie, and the rest of the province.

ELIGIBILITY:
Inclusion Criteria:

* Men >30 years of age
* Women > 40 years of age
* History of vascular disease (as defined in Study Design, page 8)
* Framingham Risk Score >/= 12 %
* Capable of giving informed consent
* Ability and willingness to complete questionnaires and have study procedures done
* Willingness to belong to either the intervention or standard care arm

Exclusion Criteria:

* FRS <12% (low risk) -- enrolled into the cohort arm (not randomized. Follow-up at study end only.)
* Any condition that will prevent the patient from participating in and completing the study
* Unable to come to the Group Health Centre for appointments
* Any factor likely to limit protocol compliance
* Unwilling to permit VIP staff to contact their primary physicians to communicate information about the study and the participant's data and treatment assignment
* Previous randomization into this study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who attained a significant reduction in their global cardiovascular risk at 6 and 12 months. This was determined a priori by the investigators to be an increase in the ACTION Score of 5 or more. | 6 months and 12 months

SECONDARY OUTCOMES:
Secondary outcomes were change in the average ACTION Score, change in individual risk domains as measured by the ACTION Score, patient satisfaction, and quality of life, all after 6 months and 12 months, comparing intervention versus control. | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Crookston, MD CCFP, Principal Investigator — Algoma District Medical Group and Group Health Centre
Locations (1):
- Group Health Centre, Sault Ste. Marie, Ontario, Canada

REFERENCES:
- See also: (Group Health Centre website) — http://www.ghc.on.ca